CLINICAL TRIAL: NCT00966875
Title: A Phase 2 Dose-Ranging Study of Multiple Subcutaneous Doses of LY2439821 (an Anti-IL-17 Antibody) in Patients With Active Rheumatoid Arthritis on Concomitant DMARD Therapy
Brief Title: A Study in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12061; I1F-MC-RHAK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- 3 mg LY2439821 (bDMARD-naive population) (Experimental): 3 milligrams (mg) LY2439821 at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60. [Biologic Disease Modifying Anti-Rheumatic Drug (bDMARD)]
  Interventions: Biological: LY2439821
- 10 mg LY2439821 (bDMARD-naive population) (Experimental): 10 mg LY2439821 at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
  Interventions: Biological: LY2439821
- 30 mg LY2439821 (bDMARD-naive population) (Experimental): 30 mg LY2439821 at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
  Interventions: Biological: LY2439821
- 80 mg LY2439821 (bDMARD-naive population) (Experimental): 80 mg LY2439821 at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
  Interventions: Biological: LY2439821
- 180 mg LY2439821 (bDMARD-naive population) (Experimental): 180 mg LY2439821 at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
  Interventions: Biological: LY2439821
- 80 mg LY2439821 (TNFa-IR population) (Experimental): 80 mg LY2439821 at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60. [Tumor Necrosis Factor Alpha-Inadequate Responder (TNFα-IR)]
  Interventions: Biological: LY2439821
- 180 mg LY2439821 (TNFa-IR population) (Experimental): 180 mg LY2439821 at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
  Interventions: Biological: LY2439821
- Placebo (bDMARD-naive population) (Placebo Comparator): Placebo at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
  Interventions: Drug: Placebo
- Placebo (TNFa-IR population) (Placebo Comparator): Placebo at Weeks 0, 1, 2, 4, 6, 8 and 10, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: LY2439821 — Subcutaneous
  Other Names: ixekizumab
  Arms: 10 mg LY2439821 (bDMARD-naive population); 180 mg LY2439821 (TNFa-IR population); 180 mg LY2439821 (bDMARD-naive population); 3 mg LY2439821 (bDMARD-naive population); 30 mg LY2439821 (bDMARD-naive population); 80 mg LY2439821 (TNFa-IR population); 80 mg LY2439821 (bDMARD-naive population)
Drug: Placebo — Subcutaneous
  Arms: Placebo (TNFa-IR population); Placebo (bDMARD-naive population)

SUMMARY:
The primary purpose of the study is to help answer the following research questions, and not to provide treatment for Rheumatoid Arthritis (RA):

* The safety of LY2439821 and any side effects that might be associated with it.
* Whether LY2439821 can help participants with active RA.
* How much LY2439821 should be given to participants.

DETAILED DESCRIPTION:
Study I1F-MC-RHAK is a multicenter study in participants with active RA on concomitant conventional DMARD therapy. The study is a Phase 2 study with 2 parts. Part A is a randomized, double-blind, placebo-controlled, parallel-group, dose-ranging design and Part B is an optional, open-label extension design. Two participant populations will be evaluated in this study: bDMARD-naive participants and TNFα-IR participants. Participants in Part A receive multiple subcutaneous injections of LY2439821 [bDMARD-naive participants: 0 (placebo), 3, 10, 30, 80, or 180 mg; TNFα-IR participants: 0 (placebo), 80 or 180 mg] at Weeks 0, 1, 2, 4, 6, 8, and 10. Participants in Part B receive subcutaneous injections of LY2439821 160 mg at Weeks 16, 18, and 20, and every 4 weeks thereafter through Week 60. Participants who complete both Part A and B have a total study participation of up to approximately 72 to 84 weeks.

ELIGIBILITY:
Inclusion Criteria:

* You must be between the ages of 18 and 75
* You must have active RA

Qualifications Specific to the bDMARD-naive Population:

You must be regularly using methotrexate (MTX) for at least 12 weeks before your participation in this study

Qualifications Specific to the TNFα-IR Population:

* You must have been treated with at least 1 biologic TNFα inhibitor therapy and either had an insufficient response to at least 3 months of treatment OR have been intolerant of such treatment
* You must be regularly using at least 1 conventional DMARD in a stable treatment regimen

Exclusion Criteria:

* You are concomitantly using non-steroidal anti-inflammatory drugs (NSAIDS), unless you are on a stable dose within the last 2 weeks
* You are a woman who is lactating or breast feeding
* You have donated more than 300 milliliters (mL) of blood within the last month
* You have received glucocorticoid administered by intra-articular, intramuscular, or intravenous injection or oral corticosteroids at an average daily dose of greater than 10 mg per day of prednisone or its equivalent within the last 4 weeks
* You had surgery on a joint that is to be assessed in the study within 2 months of study enrollment, or will require such during the study
* You have another serious disorder or illness
* You suffered a serious bacterial infection (for example, pneumonia, cellulitis, or bone or joint infections) within the last 3 months
* You have a history of uncontrolled high blood pressure
* You have clinical laboratory test results at entry that are outside the normal reference range
* You are an employee of the clinic or you are an immediate family member of an employee of the clinic. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* You are currently participating in or were discontinued within the last 30 days from another clinical trial involving an investigational drug
* If you are a woman and you could become pregnant during this study, you must talk to the study doctor about the birth control that you will use to avoid getting pregnant during the study.
* If you are a post-menopausal woman, you must be at least 45 years of age and have not menstruated for the last 12 months
* If you are a post-menopausal woman between 40 and 45 years of age, test negative for pregnancy, and have not menstruated during the last 12 months only, you must have an additional blood test to see if you can participate.
* If you are male, you must agree to reduce the risk of your female partner becoming pregnant during the study.

Exclusions Specific to the bDMARD-naive Population:

* You have received any prior bDMARD therapy such as TNFα, Interleukin (IL)-1, IL-6, T-cell, or B-cell targeted therapies
* You have had an inadequate response to a minimum of 3 months of treatment with 5 or more conventional DMARDs [such as leflunomide, azathioprine, cyclosporine, etcetera (etc.)]
* You have used DMARDs other than MTX, hydroxychloroquine, or sulfasalazine within the last 8 weeks
* You have used leflunomide within the last 12 weeks and have not received cholestyramine to speed up the elimination of leflunomide from your body.

Exclusions Specific to the TNFα-IR Population:

* You are currently using or recently used a bDMARD or a biologic TNFα inhibitor therapy within specified periods
* You have had a serious reaction to other biologic DMARDs that, in the study doctor's opinion, puts you at serious risk
* You have used cyclosporine or any other immunosuppressive in the 8 weeks before your participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (74):
- United States (37):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Desert, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Jose, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stanford, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westlake Village, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Mary, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarasota, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cumberland, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frederick, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wheaton, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bingham Farms, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sellersville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Temple, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olympia, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago, Chile
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hohenfelde
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- India (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Secunderabad
- Peru (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arequipa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pueblo Libre
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bytom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Częstochowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gmina Końskie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kościan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung County
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

REFERENCES:
- [Derived] Genovese MC, Braun DK, Erickson JS, Berclaz PY, Banerjee S, Heffernan MP, Carlier H. Safety and Efficacy of Open-label Subcutaneous Ixekizumab Treatment for 48 Weeks in a Phase II Study in Biologic-naive and TNF-IR Patients with Rheumatoid Arthritis. J Rheumatol. 2016 Feb;43(2):289-97. doi: 10.3899/jrheum.140831. Epub 2015 Dec 15. PMID 26669919
- [Derived] Genovese MC, Greenwald M, Cho CS, Berman A, Jin L, Cameron GS, Benichou O, Xie L, Braun D, Berclaz PY, Banerjee S. A phase II randomized study of subcutaneous ixekizumab, an anti-interleukin-17 monoclonal antibody, in rheumatoid arthritis patients who were naive to biologic agents or had an inadequate response to tumor necrosis factor inhibitors. Arthritis Rheumatol. 2014 Jul;66(7):1693-704. doi: 10.1002/art.38617. PMID 24623718

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to Part A and had the option of continuing in the open-label extension, Part B after completing Part A.
Groups:
- Placebo [bDMARD-naive Population]: Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 milligrams (mg) LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60. [Biologic Disease Modifying Anti-Rheumatic Drug (bDMARD)]
- 3 mg LY2439821 [bDMARD-naive Population]: 3 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 10 mg LY2439821 [bDMARD-naive Population]: 10 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 30 mg LY2439821 [bDMARD-naive Population]: 30 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 80 mg LY2439821 [bDMARD-naive Population]; 80 mg LY2439821 [TNFα-IR Population]: 80 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 180 mg LY2439821[bDMARD-naive Population]; 180 mg LY2439821 [TNFα-IR Population]: 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- Placebo [TNFα-IR Population]: Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60. [Tumor Necrosis Factor Alpha-Inadequate Responder (TNFα-IR)]
Period: Part A
Arm/Group | Placebo [bDMARD-naive Population] | 3 mg LY2439821 [bDMARD-naive Population] | 10 mg LY2439821 [bDMARD-naive Population] | 30 mg LY2439821 [bDMARD-naive Population] | 80 mg LY2439821 [bDMARD-naive Population] | 180 mg LY2439821[bDMARD-naive Population] | Placebo [TNFα-IR Population] | 80 mg LY2439821 [TNFα-IR Population] | 180 mg LY2439821 [TNFα-IR Population]
Started | 54 | 40 | 35 | 37 | 57 | 37 | 64 | 65 | 59
Received ≥1 Doses of Study Drug | 54 | 40 | 35 | 37 | 57 | 37 | 64 | 65 | 59
Completed | 48 | 36 | 33 | 34 | 52 | 33 | 52 | 58 | 51
Not Completed | 6 | 4 | 2 | 3 | 5 | 4 | 12 | 7 | 8
Not completed — Adverse Event | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 3
Not completed — Entry Criteria | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Parent/Caregiver Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Not completed — Sponsor Decision | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 1 | 3 | 0 | 5 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Period: Part B
Arm/Group | Placebo [bDMARD-naive Population] | 3 mg LY2439821 [bDMARD-naive Population] | 10 mg LY2439821 [bDMARD-naive Population] | 30 mg LY2439821 [bDMARD-naive Population] | 80 mg LY2439821 [bDMARD-naive Population] | 180 mg LY2439821[bDMARD-naive Population] | Placebo [TNFα-IR Population] | 80 mg LY2439821 [TNFα-IR Population] | 180 mg LY2439821 [TNFα-IR Population]
Started | 46 (Two (2) participants who completed Part A did not enter Part B.) | 36 | 33 | 34 | 51 (One (1) participant who completed Part A did not enter Part B.) | 32 (One (1) participant who completed Part A did not enter Part B.) | 51 (One (1) participant who completed Part A did not enter Part B.) | 57 (One (1) participant who completed Part A did not enter Part B.) | 50 (One (1) participant who completed Part A did not enter Part B.)
Completed | 41 | 33 | 27 | 31 | 44 | 26 | 29 | 38 | 32
Not Completed | 5 | 3 | 6 | 3 | 7 | 6 | 22 | 19 | 18
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 1 | 0 | 5 | 2 | 2
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 1 | 1 | 1 | 2 | 3 | 12 | 9 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 2
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 1 | 2 | 1 | 4 | 5 | 5
Not completed — Entry Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo [bDMARD-naive Population]; Placebo [TNFα-IR Population]: Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 30 mg LY2439821 [bDMARD-naive Population: 30 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- Total: Total of all reporting groups
Arm/Group | Placebo [bDMARD-naive Population] | 3 mg LY2439821 [bDMARD-naive Population] | 10 mg LY2439821 [bDMARD-naive Population] | 30 mg LY2439821 [bDMARD-naive Population | 80 mg LY2439821 [bDMARD-naive Population] | 180 mg LY2439821[bDMARD-naive Population] | Placebo [TNFα-IR Population] | 80 mg LY2439821 [TNFα-IR Population] | 180 mg LY2439821 [TNFα-IR Population] | Total
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 57 | 37 | 64 | 65 | 59 | 448
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 37 | 30 | 29 | 48 | 32 | 59 | 55 | 52 | 387
  >=65 years | 9 | 3 | 5 | 8 | 9 | 5 | 5 | 10 | 7 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.99 (10.18) | 52.19 (9.67) | 53.86 (10.62) | 53.03 (12.16) | 52.60 (10.91) | 52.21 (11.33) | 53.19 (10.44) | 54.74 (11.12) | 52.43 (9.90) | 53.08 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 33 | 27 | 31 | 52 | 30 | 55 | 57 | 51 | 383
  Male | 7 | 7 | 8 | 6 | 5 | 7 | 9 | 8 | 8 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 8 | 7 | 10 | 6 | 15 | 23 | 15 | 100
  Not Hispanic or Latino | 45 | 32 | 24 | 29 | 46 | 30 | 48 | 41 | 43 | 338
  Unknown or Not Reported | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 1 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 2 | 1 | 2 | 4 | 0 | 0 | 2 | 16
  Asian | 16 | 13 | 10 | 12 | 17 | 10 | 3 | 4 | 3 | 88
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 0 | 1 | 3 | 1 | 6 | 2 | 4 | 23
  White | 29 | 20 | 21 | 20 | 31 | 22 | 54 | 58 | 50 | 305
  More than one race | 3 | 2 | 2 | 3 | 4 | 0 | 1 | 1 | 0 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 8 | 8 | 12 | 9 | 33 | 32 | 31 | 154
  Taiwan | 5 | 4 | 3 | 4 | 4 | 3 | 1 | 1 | 1 | 26
  Argentina | 1 | 0 | 0 | 1 | 1 | 0 | 10 | 11 | 10 | 34
  Poland | 11 | 8 | 8 | 7 | 9 | 7 | 11 | 11 | 10 | 82
  Romania | 5 | 4 | 3 | 4 | 6 | 3 | 1 | 1 | 0 | 27
  Peru | 6 | 4 | 4 | 4 | 6 | 4 | 1 | 1 | 1 | 31
  Chile | 0 | 1 | 2 | 0 | 2 | 2 | 1 | 2 | 1 | 11
  Russian Federation | 3 | 1 | 0 | 1 | 3 | 2 | 1 | 1 | 1 | 13
  Germany | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 8
  Korea, Republic of | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 3 | 2 | 16
  India | 9 | 7 | 6 | 7 | 11 | 6 | 0 | 0 | 0 | 46

OUTCOME MEASURES:

1. Primary Outcome: Dose-Response Relationship Measured by the Percentage of Participants With American College of Rheumatology (ACR) 20 Response in bDMARD-Naive Population
Description: ACR20 responders are participants with at least 20% improvement from baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: Health Assessment Questionnaire-Disability Index (HAQ-DI) which measured participants perceived degree of difficulty performing daily activities, C-reactive Protein (CRP), Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), Patient's Global Assessment of Disease Activity-VAS(PtGADA-VAS), and Physician's Global Assessment of Disease Activity-VAS (PhGA-VAS). Missing values were imputed using Non-Responder Imputation (NRI). Percentage of participants achieving ACR20 response was calculated as: (number of ACR20 responders / number of participants treated) * 100.
Time Frame: Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug and were bDMARD-naive.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (bDMARD-naive Population): Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- 3 mg LY2439821 (bDMARD-naive Population): 3 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- 10 mg LY2439821 (bDMARD-naive Population): 10 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- 30 mg LY2439821 (bDMARD-naive Population): 30 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- 80 mg LY2439821 (bDMARD-naive Population): 80 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- 180 mg LY2439821 (bDMARD-naive Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 57 | 37
percentage of participants | 34.1 | 46.2 | 52.2 | 55.0 | 55.3 | 54.0
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.031, Regression, Logistic — A log transformed dose was used in the model

2. Secondary Outcome: Percentage of Participants With ACR20 Response in Tumor Necrosis Factor Alpha-Inadequate Responder (TNFα-IR) Population
Description: ACR20 responders were participants with at least 20% improvement from baseline for TJC, SJC, and at least 3 of the 5 remaining core set measures: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, and PhGA-VAS. Missing values were imputed using NRI. Percentage of participants achieving ACR20 response was calculated as: (number of ACR20 responders / number of participants treated) * 100.
Time Frame: Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug and were TNFα-IR.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (TNFα-IR Population): Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- 80 mg LY2439821 (TNFα-IR Population): 80 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- 180 mg LY2439821 (TNFα-IR Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
Arm/Group | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 64 | 65 | 59
percentage of participants | 23.4 | 40.0 | 39.0
Statistical Analysis 1: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.033, Fisher Exact
Statistical Analysis 2: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.047, Fisher Exact

3. Secondary Outcome: Smallest Doses That Achieve 10%, 50%, and 90% of the Maximum ACR 20 Response in bDMARD-Naive Population
Description: ACR20 responders are participants with at least 20% improvement from baseline for TJC, SJC, and at least 3 of the 5 remaining core set measures: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, and PhGA-VAS. The model used in the dose response analysis was used to estimate the doses that achieved 10%, 50%, and 90% of the maximal drug efficacy. Missing values were imputed using NRI. The log transformed dose was evaluated.
Time Frame: Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug and were bDMARD-naive.
Measure: Number; unit: log (dose) mg
Groups:
- 3 mg to 180 mg LY2439821 (bDMARD-naive Population): 3 mg to 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
Arm/Group | 3 mg to 180 mg LY2439821 (bDMARD-naive Population)
Number analyzed (Participants) | 206
log (dose) mg
  Estimated dose to achieve 10% response | 0.8
  Estimated dose to achieve 50% response | 2.4
  Estimated dose to achieve 90% response | 13.8

4. Secondary Outcome: Smallest Doses That Achieved 10%, 50%, and 90% of the Maximum Disease Activity Score (DAS) 28 Response in bDMARD-Naive Population
Description: DAS modified included the 28 diarthrodial joint count (DAS28) that consisted of a composite score of the following variables: TJC out of 28 (TJC28), SJC out of 28 (SJC28), CRP [milligrams per liter (mg/L)], and PtGADA on a 0 to 100 millimeter (mm) VAS ranging from 0 mm (no arthritis activity) to 100 mm (extremely active arthritis). DAS28 was calculated as: DAS28 - CRP = 0.56(square root of TJC28) + 0.28(square root of SJC28) + 0.36(ln[CRP +1]) + 0.014(VAS) + 0.96.
Time Frame: Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug and were bDMARD-naive.
Measure: Number; unit: log (dose) mg
Groups:
- 3 mg to 180 mg (bDMARD-naive Population): 3 mg to 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
Arm/Group | 3 mg to 180 mg (bDMARD-naive Population)
Number analyzed (Participants) | 206
log (dose) mg
  Estimated dose to achieve 10% response | 7.3
  Estimated dose to achieve 50 % response | 41.5
  Estimated dose to achieve 90% response | 97.0

5. Secondary Outcome: Smallest Doses That Achieve 10%, 50%, and 90% of the Maximum ACR50 Response in bDMARD-Naive Population
Description: ACR50 responders were participants with at least 50% improvement from baseline for TJC, SJC, and at least 3 of the 5 remaining core set measures: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, and PhGA-VAS. Missing values were imputed using NRI.
Time Frame: Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug and were bDMARD-naive.
Measure: Number; unit: log (dose) mg
Groups:
- 3 mg to 180 mg LY2439821 (bDMARD-naive Population): 3 mg to 180 mg LY2439821administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
Arm/Group | 3 mg to 180 mg LY2439821 (bDMARD-naive Population)
Number analyzed (Participants) | 206
log (dose) mg
  Estimated dose to achieve 10% response | 7.3
  Estimated dose to achieve 50% response | 37.9
  Estimated dose to achieve 90% response | 81.2

6. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28)-Part A
Description: DAS28 consisted of a composite score of the following variables: TJC28, SJC28, CRP, and PtGADA-VAS. DAS28 was calculated as: DAS28 - CRP =0.56(square root TJC28) + 0.28(square root SJC28) + 0.36(ln[CRP +1]) + 0.014(VAS) + 0.96. A negative change indicated an improvement.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 57 | 37 | 64 | 65 | 59
units on a scale | -0.818 (0.981) | -1.308 (1.092) | -1.565 (1.440) | -1.671 (1.193) | -1.686 (1.344) | -1.940 (1.152) | -0.619 (1.109) | -1.310 (1.303) | -1.571 (1.261)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.013, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

7. Secondary Outcome: Change From Baseline in DAS28 - Part B
Description: as for outcome 6
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 DAS28 results.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo/160 mg LY2439821 (bDMARD-naive Population); Placebo/160 mg LY2439821(TNFα-IR Population): Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 3 mg/160 mg LY2439821(bDMARD-naive Population): 3 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 10 mg/160 mg LY2439821(bDMARD-naive Population): 10 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 30 mg/160 mg LY2439821(bDMARD-naive Population): 30 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 80 mg/160 mg LY2439821(bDMARD-naive Population); 80 mg/160 mg LY2439821(TNFα-IR Population): 80 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 180 mg/160 mg LY2439821 (bDMARD-naive Population); 180 mg/160 mg LY2439821(TNFα-IR Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821(bDMARD-naive Population) | 10 mg/160 mg LY2439821(bDMARD-naive Population) | 30 mg/160 mg LY2439821(bDMARD-naive Population) | 80 mg/160 mg LY2439821(bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821(TNFα-IR Population) | 80 mg/160 mg LY2439821(TNFα-IR Population) | 180 mg/160 mg LY2439821(TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 31 | 41 | 33
units on a scale | -2.143 (1.177) | -1.832 (1.031) | -2.320 (1.292) | -2.277 (1.337) | -2.280 (1.316) | -2.475 (1.140) | -1.740 (1.460) | -1.604 (1.282) | -1.874 (1.279)

8. Secondary Outcome: Percentage of Participants With ACR20/50/70 Response - Part A
Description: ACR20 (or ACR50 or ACR70) responders were participants with at least 20% (or 50% or 70%, respectively) improvement from baseline TJC, SJC, and at least 3 of the 5 remaining core set measures: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, and PhGA-VAS. Missing values were imputed using NRI. Percentage of participants was calculated as: (number of ACR20 [or ACR50 or ACR70] responders per treatment arm) / (total number of participants per treatment arm) * 100.
Time Frame: Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 57 | 37 | 64 | 65 | 59
percentage of participants
  ACR20 | 35.2 | 45.0 | 42.9 | 70.3 | 50.9 | 54.1 | 23.4 | 40.0 | 39.0
  ACR50 | 9.3 | 17.5 | 28.6 | 29.7 | 26.3 | 27.0 | 7.8 | 20.0 | 16.9
  ACR70 | 1.9 | 5.0 | 14.3 | 13.5 | 7.0 | 13.5 | 3.1 | 3.1 | 10.2
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.227, Fisher Exact — P-value is for ACR20-NRI at Week 12
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.306, Fisher Exact — P-value is for ACR20-NRI at Week 12
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.001, Fisher Exact — P-value is for ACR20-NRI at Week 12
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.070, Fisher Exact — P-value is for ACR20-NRI at Week 12
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.058, Fisher Exact — P-value is for ACR20-NRI at Week 12
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.033, Fisher Exact — P-value is for ACR20-NRI at Week 12
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.047, Fisher Exact — P-value is for ACR20-NRI at Week 12
Statistical Analysis 8: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.191, Fisher Exact — P-value is for ACR50-NRI at Week 12
Statistical Analysis 9: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.019, Fisher Exact — P-value is for ACR50-NRI at Week 12
Statistical Analysis 10: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.013, Fisher Exact — P-value is for ACR50-NRI at Week 12
Statistical Analysis 11: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.017, Fisher Exact — P-value is for ACR50-NRI at Week 12
Statistical Analysis 12: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.026, Fisher Exact — P-value is for ACR50-NRI at Week 12
Statistical Analysis 13: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.039, Fisher Exact — P-value is for ACR50-NRI at Week 12
Statistical Analysis 14: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.102, Fisher Exact — P-value is for ACR50-NRI at Week 12
Statistical Analysis 15: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.388, Fisher Exact — P-value is for ACR70-NRI at Week 12
Statistical Analysis 16: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.033, Fisher Exact — P-value is for ACR70-NRI at Week 12
Statistical Analysis 17: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.039, Fisher Exact — P-value is for ACR70-NRI at Week 12
Statistical Analysis 18: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.199, Fisher Exact — P-value is for ACR70-NRI at Week 12
Statistical Analysis 19: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.039, Fisher Exact — P-value is for ACR70-NRI at Week 12
Statistical Analysis 20: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.696, Fisher Exact — P-value is for ACR70-NRI at Week 12
Statistical Analysis 21: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.112, Fisher Exact — P-value is for ACR70-NRI at Week 12

9. Secondary Outcome: Percentage of Participants With of ACR20/50/70 Response - Part B
Description: ACR20 (or ACR50 or ACR70) responders were participants with at least 20% (or 50% or 70% respectively) improvement from baseline TJC, SJC, and at least 3 of the 5 remaining core set measures: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, and PhGA-VAS. Missing values were imputed using NRI. Percentage of participants was calculated as: (number of ACR20 [or ACR50 or ACR70] responders per treatment arm) / (total number of participants per treatment arm) * 100].
Time Frame: Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 ACR20/50/70 results.
Measure: Number; unit: percentage of participants
Groups:
- Placebo/160 mg LY2439821(bDMARD-naive Population); Placebo/160 mg LY2439821(TNFα-IR Population): Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 3 mg/160 mg LY2439821 (bDMARD-naive Population): 3 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 10 mg/160 mg LY2439821 (bDMARD-naive Population): 10 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 30 mg/160 mg LY2439821 (bDMARD-naive Population): 30 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 80 mg/160 mg LY2439821 (bDMARD-naive Population); 80 mg/160 mg LY2439821 (TNFα-IR Population): 80 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 180 mg/160 mg LY2439821 (TNFα-IR Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
Arm/Group | Placebo/160 mg LY2439821(bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821(TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 40 | 32 | 28 | 31 | 44 | 26 | 31 | 41 | 34
percentage of participants
  ACR20 | 75.0 | 65.6 | 67.9 | 80.6 | 72.7 | 80.8 | 51.6 | 43.9 | 64.7
  ACR50 | 42.5 | 37.5 | 50.0 | 48.4 | 47.7 | 61.5 | 32.3 | 22.0 | 38.2
  ACR70 | 17.5 | 12.5 | 32.1 | 22.6 | 11.4 | 30.8 | 19.4 | 9.8 | 17.6

10. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set-TJC - Part A
Description: TJC was determined by examination of 28 joint counts that were assessed for tenderness by pressure and joint manipulation on physical examination. The participant was asked for pain sensations on these manipulations and was watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-non-tender dichotomy. Joint assessments for each participant were performed by the same assessor, when possible, throughout the study to minimize variation. Replaced, ankylosed, arthrodesed joints were identified by the investigator and excluded from evaluation during the study. Any joints that required intra-articular injections during the study were excluded from evaluation from the time of the injection to the conclusion of the study. The number of tender joints ranged from 0-28. A negative change indicated fewer tender joints.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Mean (Standard Deviation); unit: tender joints
Groups:
- 3 mg LY2439821 (bDMARD-naive Population): 3 milligram (mg) LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 56 | 37 | 64 | 65 | 59
tender joints | -2.95 (5.20) | -6.02 (7.35) | -6.79 (7.67) | -7.05 (6.28) | -7.66 (8.96) | -8.96 (7.47) | -2.96 (6.31) | -6.02 (7.31) | -6.02 (6.74)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.017, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.042, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.008, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.007, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

11. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set-TJC - Part B
Description: as for outcome 10
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 TJC results.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Placebo/160 mg LY2439821(bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821(TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 31 | 41 | 34
tender joints | -8.73 (6.85) | -8.78 (5.32) | -11.43 (6.54) | -9.55 (6.20) | -10.86 (7.48) | -10.55 (7.11) | -6.62 (8.39) | -7.35 (6.83) | -6.81 (6.11)

12. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set-SJC - Part A
Description: SJC was determined by examination of 28 joint that were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. Swelling secondary to osteoarthrosis was assessed as not swollen, unless there was unmistakable fluctuation. Joint assessments for each participant were performed by the same assessor, when possible, throughout the study to minimize variation. Replaced, ankylosed, or arthrodesed joints were identified by the investigator and were excluded from evaluation during the study. Any joints that required intra-articular injections over the course of the study were excluded from evaluation from the time of the injection to the conclusion of the study. The number of swollen joints count ranged from 0-28. A negative change indicated fewer swollen joints.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 56 | 37 | 64 | 65 | 59
swollen joints | -2.69 (6.07) | -4.25 (5.58) | -6.51 (7.65) | -6.16 (6.44) | -7.49 (7.98) | -6.52 (6.62) | -1.69 (5.93) | -5.57 (5.51) | -5.15 (5.65)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.093, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.023, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.006, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.028, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

13. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set-SJC - Part B
Description: SJC was determined by examination of 28 joint that were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint. Swelling secondary to osteoarthrosis was assessed as not swollen, unless there was unmistakable fluctuation. Joint assessments for each participant were performed by the same assessor, when possible, throughout the study to minimize variation. Replaced, ankylosed, or arthrodesed joints were identified by the investigator and were excluded from evaluation during the study. Any joints that required intra-articular injections over the course of the study were excluded from evaluation from the time of the injection to the conclusion of the study. The number of swollen joints ranged from 0-28. A negative change indicated fewer swollen joints.
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 SJC results.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo/160 mg LY2439821(bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821(TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 31 | 41 | 34
swollen joints | -7.25 (6.15) | -5.73 (4.95) | -9.06 (5.92) | -7.26 (5.73) | -8.95 (6.64) | -8.96 (6.06) | -7.32 (6.45) | -5.46 (6.51) | -6.29 (5.75)

14. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set-PAAP VAS - Part A
Description: Participants were asked to assess his/her current level of arthritis pain by marking a vertical tick on a 100-mm horizontal VAS with the left end (0 mm) marked as "no pain" and the right end (100 mm) marked "worst possible pain." The scale was administered prior to the TJC and SJC count examinations. Results were expressed in mm measured between the left end of the scale and the crossing point of the vertical line of the tick. A negative change indicated a lessening of the participant's arthritis pain.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 56 | 37 | 63 | 65 | 56
mm | -14.8 (23.7) | -18.7 (22.8) | -21.3 (28.4) | -29.8 (24.1) | -25.8 (23.0) | -25.3 (27.5) | -9.4 (24.0) | -10.3 (24.7) | -18.8 (26.6)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.247, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.315, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.006, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.042, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.055, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.365, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.005, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

15. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set-PAAP-VAS - Part B
Description: Participants were asked to assess his/her current level of arthritis pain by marking a vertical tick on a 100-mm horizontal VAS with the left end (0 mm) marked as "no pain" and the right end (100 mm) marked "worst possible pain". The scale was administered prior to the TJC and SJC count examinations. Results were expressed in mm measured between the left end of the scale and the crossing point of the vertical line of the tick. A negative change indicated a lessening of the participant's arthritis pain.
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 PAAP-VAS results.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Placebo/160 mg LY2439821 (TNFα-IR Population): Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821 (TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 31 | 41 | 34
mm | -32.5 (27.8) | -26.2 (20.3) | -33.3 (33.4) | -36.2 (27.4) | -32.4 (22.6) | -41.2 (23.0) | -25.5 (22.3) | -16.5 (21.1) | -26.2 (26.2)

16. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set - PtGADA-VAS - Part A
Description: The participant was asked to give an overall assessment of his/her current arthritis disease activity. The participants response was recorded by marking a vertical tick on a 100-mm VAS with the left end (0 mm) marked as "no arthritis activity" to the right end (100 mm) marked "extremely active arthritis." A negative change indicated an improvement in the participant's assessment of disease activity.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 56 | 37 | 63 | 65 | 58
mm | -19.2 (21.4) | -17.3 (20.9) | -18.5 (28.7) | -29.1 (23.1) | -22.1 (23.7) | -30.1 (26.9) | -10.1 (24.7) | -12.1 (27.9) | -21.6 (25.4)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.778, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.865, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.030, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.331, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.039, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.292, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.003, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

17. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set - PtGADA-VAS - Part B
Description: as for outcome 16
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 PtGADA-VAS results.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821 (TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 32 | 28 | 31 | 44 | 26 | 31 | 41 | 33
mm | -35.4 (26.2) | -24.9 (25.4) | -31.8 (30.4) | -34.8 (27.0) | -28.5 (24.7) | -39.8 (25.5) | -22.4 (23.2) | -17.8 (21.4) | -25.1 (23.9)

18. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set - PhGA-VAS - Part A
Description: The investigator gave an overall assessment of the severity of the participants disease activity. The physician's response was recorded by marking a vertical tick on a 100-mm VAS with the left end (0 mm) marked as "no arthritis activity" and the right end (100 mm) marked as "extremely active arthritis." A negative change indicated a lessening in the severity of the participant's disease activity.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 56 | 37 | 64 | 65 | 59
mm | -16.0 (19.0) | -21.0 (15.6) | -21.7 (25.2) | -26.7 (18.1) | -24.5 (22.3) | -28.8 (24.2) | -8.6 (21.4) | -25.7 (22.2) | -22.0 (24.0)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.090, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.131, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.008, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.013, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.010, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

19. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set - PhGA-VAS - Part B
Description: The investigator gave an overall assessment of the severity of the participant's disease activity. The physician's response was recorded by marking a vertical tick on a 100-mm VAS with the left end (0 mm) marked as "no arthritis activity" and the right end (100 mm) marked as "extremely active arthritis." A negative change indicated a lessening in the severity of the participant's disease activity.
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 PhGA-VAS results.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821 (TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 31 | 41 | 34
mm | -36.1 (21.7) | -30.1 (22.0) | -38.5 (28.4) | -38.0 (18.5) | -31.0 (20.7) | -44.4 (17.7) | -30.1 (22.5) | -28.9 (25.8) | -32.7 (25.2)

20. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set - CRP - Part A
Description: CRP is a biological marker of disease activity. A negative change indicated an improvement in participant's disease activity.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 56 | 37 | 64 | 65 | 59
mg/L | -1.575 (22.336) | -6.079 (10.289) | -9.435 (23.148) | -7.999 (14.740) | -11.968 (19.792) | -13.575 (25.692) | 1.229 (14.811) | -9.521 (20.312) | -8.297 (21.955)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.012, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

21. Secondary Outcome: Change From Baseline in Individual Components of the ACR Core Set - CRP - Part B
Description: as for outcome 20
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 CRP results.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821 (TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 30 | 40 | 34
mg/L | -10.548 (18.555) | -4.556 (12.937) | -11.340 (23.347) | -7.865 (22.607) | -14.519 (19.260) | -6.860 (16.745) | -12.094 (28.917) | -10.130 (18.030) | -9.004 (19.698)

22. Secondary Outcome: Percentage of Participants in European League Against Rheumatism Responder Index (EULAR) 28 - Part A
Description: Assessment of participant's rheumatoid arthritis (RA) by the EULAR that is based on the DAS 28 joint count. Participants were categorized as non-responders or responders (moderate responders + good responders). Percentage of participants was calculated as: (number of responders / number of participants) * 100.
Time Frame: Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Number; unit: percentage of participants
Groups:
- 180 mg LY2439821 (bDMARD-naive Population]); 180 mg LY2439821 (TNFα-IR Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population]) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 56 | 37 | 63 | 65 | 58
percentage of participants | 44.4 | 67.5 | 60.0 | 75.7 | 73.2 | 75.7 | 36.5 | 60.0 | 65.5
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.013, Fisher Exact — P-value is for Week 12 LOCF
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.076, Fisher Exact — P-value is for Week 12 LOCF
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.002, Fisher Exact — P-value is for Week 12 LOCF
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Week 12 LOCF
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821 (bDMARD-naive Population]); Test type: Superiority or Other; p = 0.002, Fisher Exact — P-value is for Week 12
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.006, Fisher Exact — P-value is for Week 12 LOCF
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.001, Fisher Exact — P-value is for Week 12

23. Secondary Outcome: Percentage of Participants in EULAR28 - Part B
Description: Assessment of participant's RA by the EULAR that is based on the DAS28 joint count. Participants were categorized as non-responders or responders (moderate responders + good responders). Percentage of participants was calculated as: (number of responders / number of participants) * 100.
Time Frame: Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 EULAR28 results.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821 (TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 31 | 41 | 33
percentage of participants | 90.2 | 81.8 | 82.1 | 83.9 | 84.1 | 88.5 | 64.5 | 73.2 | 69.7

24. Secondary Outcome: ACR-N - Part A
Description: ACR-N was a continuous measure of clinical, laboratory and functional outcomes in RA that characterized the percentage of improvement in RA disease activity from baseline. The index was defined as the lowest of either: the percent change in TJC, the percent change in SJC, or the median percent change of the remaining 5 ACR core criteria: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, and PhGA-VAS. For each criterion, percent change was calculated as: [(post baseline value - baseline value) / baseline value] * 100.
Time Frame: Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug with results at Week 12; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 10 mg LY2439821 (bDMARD-naive Population): 10 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 180 mg LY2439821(bDMARD-naive Population); 180 mg LY2439821 (TNFα-IR Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 47 | 36 | 34 | 36 | 54 | 35 | 56 | 60 | 54
units on a scale | -11.034 (104.809) | -0.699 (139786) | 15.162 (51.130) | 11.137 (128.516) | 18.351 (41.493) | 23.375 (42.173) | -7.356 (45.724) | 2.264 (59.277) | 11.541 (49.358)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.307, ANCOVA — P-value is for Week 12
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.104, ANCOVA — P-value is for Week 12
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.139, ANCOVA — P-value is for Week 12
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.056, ANCOVA — P-value is for Week 12
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821(bDMARD-naive Population); Test type: Superiority or Other; p = 0.048, ANCOVA — P-value is for Week 12
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.160, ANCOVA — P-value is for Week 12
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.029, ANCOVA — P-value is for Week 12

25. Secondary Outcome: ACR-N - Part B
Description: ACR-N was a continuous measure of clinical, laboratory and functional outcomes in RA that characterized the percentage of improvement in RA disease activity from baseline. The index was defined as the lowest of either: the percent change in TJC, the percent change in SJC, or the median percent change of the remaining 5 ACR core criteria: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, and PhGA-VAS. For each criterion, percent change was calculated as: [(post baseline value - baseline value)/baseline value] * 100.
Time Frame: Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 ACR-N results.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 80 mg LY2439821 (bDMARD-naive Population); 80 mg LY2439821 (TNFα-IR Population): 80 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 180 mg LY2439821 (bDMARD-naive Population); 180 mg LY2439821 (TNFα-IR Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- Placebo (TNFα-IR Population): Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821 (bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 40 | 32 | 28 | 31 | 44 | 26 | 31 | 41 | 34
units on a scale | 36.839 (42.241) | 33.154 (32.439) | 39.922 (37.930) | 34.847 (69.410) | 38.996 (30.715) | 49.152 (31.544) | 22.230 (54.682) | 14.389 (45.461) | 30.891 (41.415)

26. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale - Part A
Description: The FACIT Fatigue Scale was a brief participant-reported questionnaire measure of fatigue and consisted of 13 items that assessed tiredness, weakness and difficulty conducting usual activities due to fatigue. Each question was scored on a 5-point scale from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue. For missing data, scores were prorated using the average of the other answers in the scales as long as more than 50% of the items were answered. A negative change indicated less fatigue.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: defined as all data from all randomized participants who received at least 1 dose of study drug LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 53 | 40 | 35 | 36 | 56 | 37 | 64 | 65 | 59
units on a scale | 5.566 (9.168) | 5.725 (8.706) | 6.057 (13.512) | 8.924 (9.469) | 7.250 (9.245) | 5.838 (7.946) | 4.953 (9.152) | 4.400 (8.068) | 6.627 (8.401)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.272, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.962, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.236, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.316, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821(bDMARD-naive Population); Test type: Superiority or Other; p = 0.138, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.975, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.079, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

27. Secondary Outcome: Change From Baseline in FACIT Fatigue Scale - Part B
Description: The FACIT-Fatigue Scale was a brief participant-reported questionnaire measure of fatigue and consisted of 13 items that assessed tiredness, weakness and difficulty conducting usual activities due to fatigue. Each question was scored on a 5-point scale from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue. For missing data, scores were prorated using the average of the other answers in the scales as long as more than 50% of the items were answered. A negative change indicated less fatigue.
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 FACIT results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821 (TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 31 | 41 | 34
units on a scale | 8.390 (8.405) | 4.879 (10.810) | 8.500 (12.880) | 9.177 (11.637) | 7.295 (10.436) | 6.038 (9.986) | 8.323 (9.304) | 4.341 (8.493) | 6.647 (9.639)

28. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness (Minutes) - Part A
Description: The investigator queried the participants about the duration of morning stiffness in and around their joints and the results (in minutes) were recorded by the investigator. Duration was the time from when the participants woke up to when normal activities could be resumed. Durations recorded as longer than 12 hours (720 minutes) were summarized as 720 minutes. An increase in duration from baseline indicated a joint worsening and a decrease from baseline indicated joint improvement.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 34 | 37 | 56 | 37 | 64 | 65 | 58
minutes | -36.6 (123.7) | -24.3 (87.3) | -52.7 (142.0) | -71.4 (143.9) | -63.0 (57.0) | -69.0 (64.1) | -36.3 (137.7) | -62.0 (138.1) | -43.1 (116.7)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.982, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.276, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.050, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.010, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821(bDMARD-naive Population); Test type: Superiority or Other; p = 0.046, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.017, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.066, ANCOVA — P-value is for Week 12; ANCOVA adjusted for treatment and baseline value

29. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness (Minutes) - Part B
Description: as for outcome 28
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 Duration of Morning Stiffness results.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo/160 mg LY2439821(bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821 (TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 27 | 31 | 44 | 25 | 31 | 41 | 34
minutes | -92.1 (111.3) | -70.2 (112.3) | -55.6 (72.9) | -92.3 (136.7) | -68.8 (72.5) | -82.3 (79.2) | -61.3 (161.9) | -60.9 (164.7) | -85.9 (74.8)

30. Secondary Outcome: Change From Baseline in HAQ-DI - Part A
Description: HAQ-DI was a participant-reported questionnaire that consisted of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do). The highest score for any question in a category was the score of that category unless special aids or devices or help from another person was required. Answers for at least 6 of the 8 disability domains were required to compute the participant's HAQ-DI score. If the participant had scores for fewer than 6 categories, the HAQ-DI score was considered missing. The HAQ-DI score was calculated as the sum of the category scores divided by the number of categories scored, with a possible scores range of 0 to 3. Negative mean changes from baseline indicated improvement.
Time Frame: Baseline, up to Week 12
Population: Part A FAS: All randomized participants who received at least 1 dose of study drug; LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 56 | 37 | 64 | 65 | 59
units on a scale | -0.220 (0.459) | -0.322 (0.493) | -0.418 (0.693) | -0.537 (0.639) | -0.469 (0.517) | -0.476 (0.655) | -0.182 (0.458) | -0.223 (0.448) | -0.265 (0.496)
Statistical Analysis 1: Comparison: Placebo (bDMARD-naive Population) vs 3 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.538, Fisher Exact — P-value is for Week 12
Statistical Analysis 2: Comparison: Placebo (bDMARD-naive Population) vs 10 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.515, Fisher Exact — P-value is for Week 12
Statistical Analysis 3: Comparison: Placebo (bDMARD-naive Population) vs 30 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.030, Fisher Exact — P-value is for Week 12
Statistical Analysis 4: Comparison: Placebo (bDMARD-naive Population) vs 80 mg LY2439821 (bDMARD-naive Population); Test type: Superiority or Other; p = 0.053, Fisher Exact — P-value is for Week 12
Statistical Analysis 5: Comparison: Placebo (bDMARD-naive Population) vs 180 mg LY2439821(bDMARD-naive Population); Test type: Superiority or Other; p = 0.393, Fisher Exact — P-value is for Week 12
Statistical Analysis 6: Comparison: Placebo (TNFα-IR Population) vs 80 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.077, Fisher Exact — P-value is for Week 12
Statistical Analysis 7: Comparison: Placebo (TNFα-IR Population) vs 180 mg LY2439821 (TNFα-IR Population); Test type: Superiority or Other; p = 0.105, Fisher Exact — P-value is for Week 12

31. Secondary Outcome: Change From Baseline in HAQ-DI - Part B
Description: HAQ-DI was a participant-reported questionnaire that consisted of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do). The highest score for any question in a category was the score of that category unless special aids or devices or help from another person was required. Answers for at least 6 of the 8 disability domains were required to compute the participant's HAQ-DI score. If the participant had scores for fewer than 6 categories, the HAQ-DI score was considered missing. The HAQ-DI score was calculated as the sum of the category scores divided by the number of categories scored, with a possible scores range from 0 to 3. Negative mean changes from baseline indicated improvement.
Time Frame: Baseline, Week 64
Population: All participants from Part A who entered the open-label portion of the study, Part B, with Week 64 HAQ-DI results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/160 mg LY2439821 (bDMARD-naive Population) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) | Placebo/160 mg LY2439821 (TNFα-IR Population) | 80 mg/160 mg LY2439821 (TNFα-IR Population) | 180 mg/160 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 41 | 33 | 28 | 31 | 44 | 26 | 31 | 41 | 34
units on a scale | -0.616 (0.609) | -0.542 (0.611) | -0.665 (0.662) | -0.673 (0.705) | -0.554 (0.614) | -0.697 (0.571) | -0.331 (0.449) | -0.250 (0.460) | -0.309 (0.437)

32. Secondary Outcome: Relationship Between Exposure and Response of Individual Components of the ACR Core Set
Time Frame: Through Week 72
Population: Relationship between exposure and response in Individual Components (IC) of ACR Core Set analysis was reported in outcome measures (OMs) 10-21 as change from baseline in IC of ACR Core Sets: TJC, SJC, PAAP-VAS, PtGADA-VAS, PhGA-VAS, and CRP (Parts A and B). No further analyses were completed for individual components of ACR Core Set.
Groups:
- Placebo (bDMARD-naive Population); Placebo (TNFα-IR Population): Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 3 mg LY2439821 (bDMARD-naive Population): 3 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 30 mg LY2439821 (bDMARD-naive Population): 30 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 180 mg LY2439821(bDMARD-naive Population); 180 mg LY2439821 (TNFα-IR Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Relationship Between Exposure and Response of ACR20/50/70/N
Time Frame: Through Week 72
Population: Relationship between exposure and response ACR20/50/70/N analysis was reported in OMs 8 and 9, as percentage of participants with ACR 20/50/70 Response (Parts A and B) and OMs 24 and 25 as percentage of participants with ACR-N (Parts A and B) respectively. No further analyses were completed for ACR20/50/70/N.
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Relationship Between Exposure and Response of DAS28
Time Frame: Through Week 72
Population: Relationship between exposure and response of DAS28 analysis was reported in OMs 6 and 7 as change from baseline in DAS28 (Parts A and B) respectively. No further analyses were completed for DAS28.
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Relationship Between Exposure and Response of EULAR28
Time Frame: Through Week 72
Population: Relationship between exposure and response of EULAR 28 analysis was reported in OMs 22 and 23 as percentage of participants in EULAR28 (Parts A and B), respectively. No further analyses were completed for EULAR28.
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2439821 at Steady State
Description: Evaluable PK concentrations from all time points, including data from placebo participants who elected active treatment in Part B, were combined and utilized in a population approach to determine the population median estimates and 90% confidence intervals at steady state. Day 0 and Week 6 postdose samples were collected as late as possible during the dosing visit (in other words, the postdose samples were collected at the end of their respective visits).
Time Frame: Predose: Day 0, Day 1 or 2 or 3, Day 7, Weeks 6, 10, 16, 40 and 64 and Postdose: Day 0 and Week 6
Population: All randomized participants who received at least 1 dose of study drug in Part A and had estimable PK data, as well as, participants from Part A who entered the open-label portion of the study, Part B, and had estimable PK data.
Measure: Median (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Groups:
- Part A: 3 mg LY2439821 (bDMARD-naive Population): 3 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- Part A: 10 mg LY2439821 (bDMARD-naive Population): 10 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- Part A: 30 mg LY2439821 (bDMARD-naive Population): 30 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- Part A: 80 mg LY2439821 (bDMARD-naive Population); Part A: 80 mg LY2439821 (TNFα-IR Population): 80 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- Part A: 180 mg LY2439821(bDMARD-naive Population); Part A: 180 mg LY2439821 (TNFα-IR Population): 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A.
- Part B: 160 mg LY2439821 (bDMARD-naive and TNFα-IR Population): 160 mg LY2439821 administered subcutaneously at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60, in Part B.
Arm/Group | Part A: 3 mg LY2439821 (bDMARD-naive Population) | Part A: 10 mg LY2439821 (bDMARD-naive Population) | Part A: 30 mg LY2439821 (bDMARD-naive Population) | Part A: 80 mg LY2439821 (bDMARD-naive Population) | Part A: 180 mg LY2439821(bDMARD-naive Population) | Part A: 80 mg LY2439821 (TNFα-IR Population) | Part A: 180 mg LY2439821 (TNFα-IR Population) | Part B: 160 mg LY2439821 (bDMARD-naive and TNFα-IR Population)
Number analyzed (Participants) | 40 | 35 | 37 | 57 | 37 | 65 | 59 | 390
nanograms per milliliter (ng/mL) | 336 [138 to 783] | 1060 [352 to 2580] | 3230 [1140 to 7970] | 7580 [2590 to 18600] | 17100 [6870 to 42000] | 7320 [2740 to 17700] | 16200 [6040 to 40600] | 18600 [8040 to 45000]

37. Secondary Outcome: Percentage of Participants With Anti-LY2439821 Antibodies
Description: Treatment-emergent anti-LY2439821 antibody positive participants were defined as a titer change from baseline that was at least 2 dilutions (4-fold) increase. Participants must have had an assessment to be classified as treatment emergent antibody positive or negative.
Time Frame: Week 16, Week 64
Population: Part A (Week 16) FAS: all randomized participants who received at least 1 dose of study drug with antibody testing performed; Part B (Week 64): All participants from Part A who entered the open-label portion of the study, part B, with baseline and at least 1 post-baseline antibody testing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (bDMARD-naive Population) | 3 mg LY2439821 (bDMARD-naive Population) | 10 mg LY2439821 (bDMARD-naive Population) | 30 mg LY2439821 (bDMARD-naive Population) | 80 mg LY2439821 (bDMARD-naive Population) | 180 mg LY2439821(bDMARD-naive Population) | Placebo (TNFα-IR Population) | 80 mg LY2439821 (TNFα-IR Population) | 180 mg LY2439821 (TNFα-IR Population)
Number analyzed (Participants) | 54 | 40 | 35 | 37 | 57 | 37 | 34 | 65 | 59
percentage of participants
  Part A Week 16 (n=43,35,34,35,49,33,52,57,51) | 11.6 | 14.3 | 8.8 | 8.6 | 16.3 | 15.2 | 7.7 | 10.5 | 13.7
  Part B Week 64 (n=37,32,28,30,40,26,31,41,33) | 0.0 | 0.0 | 3.6 | 0.0 | 2.5 | 3.8 | 6.5 | 0.0 | 9.1

ADVERSE EVENTS:
Groups:
- 3 mg LY2439821 (bDMARD-naive Population) Part A; 3 mg/160 mg LY2439821 (bDMARD-naive Population) Part B: 3 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 10 mg LY2439821 (bDMARD-naive Population) Part A; 10 mg/160 mg LY2439821 (bDMARD-naive Population) Part B: 10 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 30 mg LY2439821 (bDMARD-naive Population) Part A; 30 mg/160 mg LY2439821 (bDMARD-naive Population) Part B: 30 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 80 mg LY2439821 (bDMARD-naive Population) Part A; 80 mg LY2439821 (TNFa-IR Population) Part A; 80 mg/160 mg LY2439821 (bDMARD-naive Population) Part B; 80 mg/160 mg LY2439821 (TNFa-IR Population) Part B: 80 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- 180 mg LY2439821(bDMARD-naive Population) Part A; 180 mg LY2439821 (TNFa-IR Population) Part A; 180 mg/160 mg LY2439821 (bDMARD-naive Population) Part B; 180 mg/160 mg LY2439821 (TNFa-IR Population) Part B: 180 mg LY2439821 administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
- Placebo (bDMARD-naive Population) Part A; Placebo (TNFa-IR Population) Part A; Placebo/160 mg LY2439821 (bDMARD-naive Population) Part B; Placebo/160 mg LY2439821 (TNFa-IR Population) Part B: Placebo administered subcutaneously at Weeks 0, 1, 2, 4, 6, 8 and 10 in Part A, followed by 160 mg LY2439821 in Part B (optional) at Weeks 16, 18, 20 and every 4 weeks thereafter through Week 60.
Arm/Group | 3 mg LY2439821 (bDMARD-naive Population) Part A | 10 mg LY2439821 (bDMARD-naive Population) Part A | 30 mg LY2439821 (bDMARD-naive Population) Part A | 80 mg LY2439821 (bDMARD-naive Population) Part A | 180 mg LY2439821(bDMARD-naive Population) Part A | Placebo (bDMARD-naive Population) Part A | 80 mg LY2439821 (TNFa-IR Population) Part A | 180 mg LY2439821 (TNFa-IR Population) Part A | Placebo (TNFa-IR Population) Part A | 3 mg/160 mg LY2439821 (bDMARD-naive Population) Part B | 10 mg/160 mg LY2439821 (bDMARD-naive Population) Part B | 30 mg/160 mg LY2439821 (bDMARD-naive Population) Part B | 80 mg/160 mg LY2439821 (bDMARD-naive Population) Part B | 180 mg/160 mg LY2439821 (bDMARD-naive Population) Part B | Placebo/160 mg LY2439821 (bDMARD-naive Population) Part B | 80 mg/160 mg LY2439821 (TNFa-IR Population) Part B | 180 mg/160 mg LY2439821 (TNFa-IR Population) Part B | Placebo/160 mg LY2439821 (TNFa-IR Population) Part B
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/35 | 1/37 | 4/57 | 1/37 | 1/54 | 5/65 | 6/59 | 1/64 | 3/36 | 3/33 | 2/34 | 4/51 | 1/32 | 4/46 | 7/57 | 4/50 | 7/51
Other Adverse Events (participants affected / at risk) | 16/40 | 16/35 | 16/37 | 23/57 | 16/37 | 22/54 | 31/65 | 32/59 | 32/64 | 14/36 | 19/33 | 12/34 | 23/51 | 16/32 | 26/46 | 23/57 | 16/50 | 23/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 3 mg LY2439821 (bDMARD-naive Population) Part A (N=40) | 10 mg LY2439821 (bDMARD-naive Population) Part A (N=35) | 30 mg LY2439821 (bDMARD-naive Population) Part A (N=37) | 80 mg LY2439821 (bDMARD-naive Population) Part A (N=57) | 180 mg LY2439821(bDMARD-naive Population) Part A (N=37) | Placebo (bDMARD-naive Population) Part A (N=54) | 80 mg LY2439821 (TNFa-IR Population) Part A (N=65) | 180 mg LY2439821 (TNFa-IR Population) Part A (N=59) | Placebo (TNFa-IR Population) Part A (N=64) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=36) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=33) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=34) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=51) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=32) | Placebo/160 mg LY2439821 (bDMARD-naive Population) Part B (N=46) | 80 mg/160 mg LY2439821 (TNFa-IR Population) Part B (N=57) | 180 mg/160 mg LY2439821 (TNFa-IR Population) Part B (N=50) | Placebo/160 mg LY2439821 (TNFa-IR Population) Part B (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum sickness-like reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Whipple's disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/33 (0) | 0/27 (0) | 0/31 (0) | 0/52 (0) | 0/30 (0) | 0/47 (0) | 0/57 (0) | 0/51 (0) | 0/55 (0) | 0/29 (0) | 0/25 (0) | 0/29 (0) | 0/46 (0) | 0/25 (0) | 0/40 (0) | 0/49 (0) | 1/45 (1) | 0/45 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/33 (0) | 0/27 (0) | 0/31 (0) | 0/52 (0) | 0/30 (0) | 0/47 (0) | 0/57 (0) | 0/51 (0) | 0/55 (0) | 0/29 (0) | 0/25 (0) | 0/29 (0) | 0/46 (0) | 0/25 (0) | 0/40 (0) | 0/49 (0) | 1/45 (1) | 0/45 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/33 (0) | 0/27 (0) | 0/31 (0) | 0/52 (0) | 0/30 (0) | 0/47 (0) | 0/57 (0) | 1/51 (1) | 0/55 (0) | 0/29 (0) | 0/25 (0) | 0/29 (0) | 0/46 (0) | 0/25 (0) | 0/40 (0) | 0/49 (0) | 0/45 (0) | 0/45 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 3 mg LY2439821 (bDMARD-naive Population) Part A (N=40) | 10 mg LY2439821 (bDMARD-naive Population) Part A (N=35) | 30 mg LY2439821 (bDMARD-naive Population) Part A (N=37) | 80 mg LY2439821 (bDMARD-naive Population) Part A (N=57) | 180 mg LY2439821(bDMARD-naive Population) Part A (N=37) | Placebo (bDMARD-naive Population) Part A (N=54) | 80 mg LY2439821 (TNFa-IR Population) Part A (N=65) | 180 mg LY2439821 (TNFa-IR Population) Part A (N=59) | Placebo (TNFa-IR Population) Part A (N=64) | 3 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=36) | 10 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=33) | 30 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=34) | 80 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=51) | 180 mg/160 mg LY2439821 (bDMARD-naive Population) Part B (N=32) | Placebo/160 mg LY2439821 (bDMARD-naive Population) Part B (N=46) | 80 mg/160 mg LY2439821 (TNFa-IR Population) Part B (N=57) | 180 mg/160 mg LY2439821 (TNFa-IR Population) Part B (N=50) | Placebo/160 mg LY2439821 (TNFa-IR Population) Part B (N=51)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 3 (3)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (5) | 3 (3) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 5 (13) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 2 (4) | 0 (0) | 1 (4) | 3 (8) | 4 (7) | 3 (7)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (5) | 1 (3) | 6 (7) | 7 (8) | 3 (3) | 1 (6) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (14) | 0 (0) | 1 (2) | 5 (22)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (5) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (4) | 2 (3) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 3 (4) | 4 (4) | 3 (6) | 2 (2) | 3 (4) | 5 (5) | 6 (9) | 1 (1) | 1 (2)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 4 (5) | 6 (6) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (3) | 4 (5) | 4 (4) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1/33 (1) | 1/27 (1) | 0/31 (0) | 0/52 (0) | 0/30 (0) | 1/47 (1) | 0/57 (0) | 0/51 (0) | 0/55 (0) | 0/29 (0) | 0/25 (0) | 0/29 (0) | 0/46 (0) | 0/25 (0) | 2/40 (2) | 0/49 (0) | 0/45 (0) | 0/45 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 1 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 6 (7) | 7 (7) | 2 (2) | 5 (6) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 2 (3) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/7 (0) | 0/8 (0) | 0/6 (0) | 0/5 (0) | 0/7 (0) | 0/7 (0) | 0/8 (0) | 0/8 (0) | 0/9 (0) | 0/7 (0) | 0/8 (0) | 0/5 (0) | 0/5 (0) | 0/7 (0) | 1/6 (1) | 0/8 (0) | 0/5 (0) | 0/6 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (3) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (5) | 2 (2) | 2 (2) | 2 (2) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days